CLINICAL TRIAL: NCT01266460
Title: A Phase II Evaluation of ADXS11-001 (NSC 752718) in the Treatment of Persistent or Recurrent Squamous or Non-Squamous Cell Carcinoma of the Cervix
Brief Title: Vaccine Therapy in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Advaxis, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0265; NCI-2011-02671 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0265; CDR0000691288; GOG-0265 (Other: NRG Oncology); GOG-0265 (Other: CTEP); U10CA180830 (NIH); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ADXS11-001) (Experimental): Patients receive live-attenuated Listeria monocytogenes cancer vaccine ADXS11-001 IV over 30 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Attenuated Live Listeria Encoding HPV 16 E7 Vaccine ADXS11-001; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Attenuated Live Listeria Encoding HPV 16 E7 Vaccine ADXS11-001 — Given IV
  Other Names: ADXS11-001; ADXS11-001 Vaccine; Attenuated Live Listeria Encoding HPV 16 E7 Vaccine; Attenuated Live Listeria Encoding Human Papilloma Virus 16 E7 Vaccine; Lm-LLO-E7; Lovaxin-C
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well vaccine therapy works in treating patients with cervical cancer that does not go to remission despite treatment (persistent) or has come back (recurrent). Vaccines therapy may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the tolerability, safety, and nature and degree of toxicity of ADXS11-001 (live-attenuated Listeria monocytogenes cancer vaccine ADXS11-001) by the numbers of patients with dose-limiting toxicities (DLTs) and adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0.

II. To assess the activity of ADXS11-001 for patients with persistent or recurrent carcinoma of the cervix with the frequency of patients who survive for at least 12 months after initiating therapy.

SECONDARY OBJECTIVES:

I. To characterize the distribution of progression-free survival and overall survival.

II. To examine the proportion of patients with objective tumor response.

TERTIARY OBJECTIVES:

I. To assess changes in clinical immunology based upon serum cytokines and to correlate any observed changes with clinical response including progression-free survival, overall survival, tumor response, DLTs, and adverse effects.

II. To examine associations between presence and type of high-risk human papillomavirus (H-HPV) and measures of clinical response and serum cytokine levels.

OUTLINE:

Patients receive live-attenuated Listeria monocytogenes cancer vaccine ADXS11-001 intravenously (IV) over 30 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent or recurrent squamous or non-squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix with documented disease progression (disease not amenable to curative therapy); histologic confirmation of the original primary tumor is required via the pathology report
* Patient must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded)
  * Each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray
  * Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one ?target lesion? to be used to assess response on this protocol as defined by RECIST 1.1

  * Tumors within a previously irradiated field will be designated as ?non-target? lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists

  * In general, this would refer to any active GOG phase III or rare tumor protocol for the same patient population
* Patients must have a GOG performance status of 0 or 1
* Recovered from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration

  * Continuation of hormone replacement therapy is permitted
* Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted (non-cytotoxic) agents and immunologic agents, must be discontinued at least three weeks prior to registration
* Any prior radiation therapy must be completed at least 4 weeks prior to registration
* Patients must have had one prior systemic chemotherapeutic regimen for management of advanced, metastatic, or recurrent carcinoma of the cervix

  * Chemotherapy administered concurrent with primary radiation (e.g.; weekly cisplatin) is not counted as a systemic chemotherapy regimen for management of advanced, metastatic, or recurrent disease; adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is not counted as a systemic chemotherapy regimen for management of advanced, metastatic, or recurrent disease (e.g.; paclitaxel and carboplatin for up to 4 cycles)
* Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their primary therapy and/or as part of their therapy for advanced, metastatic, or recurrent disease (e.g., bevacizumab)
* Platelet count greater than or equal to 75,000/mcL
* Absolute neutrophil count (ANC) count greater than or equal to 1,000/mcL
* Lymphocyte count greater than or equal to 700/mcL
* Hemoglobin count greater than or equal to 9 g/dL or greater than or equal to 5.6 mmol/L

  * Note: ANC, platelets, hemoglobin requirement cannot be met by the use of recent transfusions, or growth factor support (granulocyte colony-stimulating factor [G-CSF], erythropoietin, etc.) within 2 weeks prior to treatment initiation
* Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN) or measured or calculated creatinine clearance greater than or equal to 50 mL/min for subject with creatinine levels greater than 1.5 x institutional ULN; (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) (creatinine clearance should be calculated per institutional standard)
* Total bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) less than or equal to 1.5 x ULN, unless patient is receiving anticoagulant therapy as long as PT or INR is within therapeutic range of intended use of anticoagulants
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements as specified
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and must agree to ongoing use of 2 methods of study doctor approved birth control or abstain from heterosexual activity for the course of the study from screening through 120 days after the last dose of study medication; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Patients cannot be lactating
* Patients must be able to swallow pills

Exclusion Criteria:

* Patients who have received prior therapy with ADXS11-001
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted below are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of cervical cancer within the last three years are excluded

  * Prior radiation for localized cancer of the breast, head and neck, or skin is permitted provided that it was completed more than three years prior to registration and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of cervical cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with a contraindication (e.g. sensitivity/allergy) to trimethoprim/sulfamethoxazole or ampicillin
* Patients allergic to nonsteroidal antiinflammatory drug (NSAID)
* Patients with active infection requiring systemic therapy or who are dependent on or currently receiving antibiotics that cannot be discontinued before dosing; (Note: subjects who discontinue an antibiotic prior to dosing must wait at least 5 half-lives after the last dose of antibiotic before receiving any ADXS11-001 infusion)
* Patients with a diagnosis of immunodeficiency, or who are dependent on or have received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment with the exception of topical corticosteroids and occasional inhaled corticosteroids, as indicated
* Patients with uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Patients with liver cirrhosis or any other impaired hepatic function as determined by serum enzymes
* Patients known to be seropositive for human immunodeficiency virus (HIV) and/or active hepatitis, even if liver function studies are in the eligible range
* Patients with a prior history of a splenectomy and/or sickle cell trait/disease
* Patient has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)); NOTE: more common devices and prosthetics which include arterial and venous stents, dental and breast implants and venous access devices (e.g., Port-a-Cath or Mediport) are permitted; sponsor must be contacted prior to consenting any subject who has any other device and/or implant
* Any patient currently requiring or anticipated to require tumor necrosis factor (TNF) blocking agent (e.g., infliximab) therapy for diagnosis of rheumatologic disease or inflammatory bowel disease (e.g., ankylosing spondylitis, Crohn disease, plaque psoriasis, psoriatic arthritis, rheumatoid arthritis or ulcerative colitis)
* Patient has undergone a major surgery, including surgery for a new artificial implant and/or device, within 6 weeks prior to the initiation of ADXS11-001 treatment; NOTE: all toxicities and/or complications must have recovered to baseline or grade 1 prior to the initiation of ADXS11-001 study therapy; sponsor must be consulted prior to enrolling patients on the study who recently had a major surgery or have new artificial implant, and/or devices
* Patient has a known allergy to any component of the study treatment formulations
* Patient has a history of listeriosis or prior ADXS11-001 therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warner K Huh, Principal Investigator — NRG Oncology
Locations (24):
- United States (24):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Huh WK, Brady WE, Fracasso PM, Dizon DS, Powell MA, Monk BJ, Leath CA 3rd, Landrum LM, Tanner EJ, Crane EK, Ueda S, McHale MT, Aghajanian C. Phase II study of axalimogene filolisbac (ADXS-HPV) for platinum-refractory cervical carcinoma: An NRG oncology/gynecologic oncology group study. Gynecol Oncol. 2020 Sep;158(3):562-569. doi: 10.1016/j.ygyno.2020.06.493. Epub 2020 Jul 6. PMID 32641240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG-0265 enrolled 54 patients from May 23, 2011 to September of 2015. Of the 54 patients enrolled, 50 patients received treatment.
Period: Overall Study
Arm/Group | Treatment (ADXS11-001)
Started | 50
Completed | 16
Not Completed | 34
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5
Not completed — Disease Progression | 18
Not completed — Not otherwise specified | 8

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 years | 25
  30 - 39 years | 11
  40 - 49 years | 17
  50 - 59 years | 9
  60 - 69 years | 10
  70 - 79 years | 1
  >= 80 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 37
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities, as Assessed by CTCAE v 4.0
Description: Number of patients with dose-limiting toxicities, as assessed by CTCAE v 4.0
Time Frame: 28 days
Population: Only the first six patients were analyzed for Dose Limiting Toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Incidence of Adverse Effects as Assessed by CTCAE v 4.0
Description: Incidence of adverse effects as assessed by CTCAE v 4.0 (i.e. the number of patients experiencing at least one grade 3 adverse event)
Time Frame: Adverse events were collected an average of 4 years 7 months
Population: Eligible and evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Participants | 29

3. Primary Outcome: Number of Patients Who Survive for at Least 12 Months
Description: The number of patients (and percentage) who survive for at least 12 months.
Time Frame: 12 months
Population: Eligible and evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Participants | 19

4. Secondary Outcome: Distribution of Overall Survival
Description: Characterized with Kaplan-Meier plots and estimates of the median time until death.
Time Frame: Patients will be followed (physical exams and histories) every three months for the first three years, then every six months for the next two years. Patients will be monitored for delayed toxicity and survival for 5-year period, unless consent withdrawn.
Population: Eligible and evaluable.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Months | 6.1 [4.3 to 12.1]

5. Secondary Outcome: Distribution of Progression-free Survival
Description: Characterized with Kaplan-Meier plots and estimates of the median time until progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 4
Population: Eligible and evaluable
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Months | 2.8 [2.6 to 3.0]

6. Secondary Outcome: Number of Patients Who Have Objective Tumor Response (Complete or Partial)
Description: The number of patients who have objective tumor response (complete response or partial response). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 4
Population: Eligible and evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ADXS11-001)
Number analyzed (Participants) | 50
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 5
  Progressive Disease | 32
  Not Evaluable | 11

7. Other Pre Specified Outcome: Changes in Clinical Immunology Based Upon Serum
Description: Examined with descriptive statistics and graphics, and their relationship with survival and tumor response will be examined with proportional hazards and logistic regression models, as appropriate.
Time Frame: Baseline to up to 24 hours after dose 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each patient, adverse events are collected from study entry until the end of follow up, an average of 4 years 7 months.
Arm/Group | Treatment (ADXS11-001)
All-Cause Mortality (participants affected / at risk) | 43/50
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (ADXS11-001) (N=50)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Alkaline phosphatase increased (Investigations) | 1
Ascites (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 1
Chills (General disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 4
Cytokine release syndrome (Immune system disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 3
Flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
GGT increased (Investigations) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
INR increased (Investigations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lethargy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Urinary tract obstruction (Renal and urinary disorders) | 3
Urine output decreased (Investigations) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (ADXS11-001) (N=50)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 14
Acute kidney injury (Renal and urinary disorders) | 4
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anal pain (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 13
Anxiety (Psychiatric disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Ascites (Gastrointestinal disorders) | 2
Aspartate aminotransferase increased (Investigations) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 17
Bladder perforation (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac troponin I increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 29
Cholecystitis (Hepatobiliary disorders) | 1
Cholesterol high (Investigations) | 1
Constipation (Gastrointestinal disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 5
Cystitis noninfective (Renal and urinary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 8
Depression (Psychiatric disorders) | 8
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Duodenal stenosis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Edema limbs (General disorders) | 13
Edema trunk (General disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Fatigue (General disorders) | 37
Fever (General disorders) | 20
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Flu like symptoms (General disorders) | 8
Flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
GGT increased (Investigations) | 14
Gallbladder pain (Hepatobiliary disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 18
Hematuria (Renal and urinary disorders) | 4
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hypotension (Vascular disorders) | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
INR increased (Investigations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 8
Localized edema (General disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphedema (Vascular disorders) | 3
Lymphocyte count decreased (Investigations) | 5
Malaise (General disorders) | 4
Memory impairment (Nervous system disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 20
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Paresthesia (Nervous system disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral nerve infection (Infections and infestations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7
Photophobia (Eye disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 11
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary frequency (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 5
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 2
Vaginal fistula (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 3
Vaginal infection (Infections and infestations) | 1
Vaginal pain (Reproductive system and breast disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 15
Weight loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT01266460/Prot_SAP_000.pdf